CLINICAL TRIAL: NCT01306591
Title: Randomized Multi-center Clinical Study：Bevacizumab for Neovascular Age-related Macular Degeneration
Brief Title: Bevacizumab for Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Peking University People's Hospital, Peking University People's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Bevacizumab for nAMD
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2010-12

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: neovascular age-related macular degeneration; Bevacizumab; Multicenter Randomized Study
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab 1 (Active Comparator)
  Interventions: Drug: Bevacizumab 1
- Bevacizumab 2 (Active Comparator)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab 1 — Bevacizumab, 1.25mg/0.05ml, every 6 weeks, 42weeks
  Arms: Bevacizumab 1
Drug: Bevacizumab — Bevacizumab, 1.25mg/0.05ml, 0week(baseline), 6week, 12week, 24week, 36week
  Arms: Bevacizumab 2

SUMMARY:
Age-related macular degeneration (AMD) is one of primary blinding eye disease among people over 65 years in China. The anti-VEGF antibody treatment is proved useful for Neovascular Age-related Macular Degeneration (nAMD) by many studies. Bevacizumab is the only available low-cost type of anti-VEGF drug currently in China. This study is a multi-center, randomized trial of Bevacizumab effective dose and safety for nAMD. This study is to explore the effective therapeutic approach that the majority of patients in China can bear establishing a suitable treatment for China.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of neovascular Age-related macular degeneration
* Signed informed consent

Exclusion Criteria:

* No other ocular fundus diseases

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
EDTRS visual acuity score | 0week(baseline), 6week, 12week, 18week, 24week, 30week, 36week, 42week, 48week
  EDTRS visual acuity score is assessed at each timepoint for every group

SECONDARY OUTCOMES:
macular thickness in OCT | 0week(baseline), 6week, 12week, 18week, 24week, 30week, 36week, 42week, 48week
  macular thickness is assessed at each timepoint for every group

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxin Li, doctor, Study Chair — Peking University People's Hospital
Locations (1):
- Xiaoxin Li, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li E, Donati S, Lindsley KB, Krzystolik MG, Virgili G. Treatment regimens for administration of anti-vascular endothelial growth factor agents for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 May 5;5(5):CD012208. doi: 10.1002/14651858.CD012208.pub2. PMID 32374423
- [Derived] Fang K, Tian J, Qing X, Li S, Hou J, Li J, Yu W, Chen D, Hu Y, Li X. Predictors of visual response to intravitreal bevacizumab for treatment of neovascular age-related macular degeneration. J Ophthalmol. 2013;2013:676049. doi: 10.1155/2013/676049. Epub 2013 Aug 28. PMID 24069533
- [Derived] Li X, Hu Y, Sun X, Zhang J, Zhang M; Neovascular Age-Related Macular Degeneration Treatment Trial Using Bevacizumab (NATTB). Bevacizumab for neovascular age-related macular degeneration in China. Ophthalmology. 2012 Oct;119(10):2087-93. doi: 10.1016/j.ophtha.2012.05.016. Epub 2012 Jul 20. PMID 22818896